CLINICAL TRIAL: NCT05957679
Title: Preoperative Evaluation of Tumor Stiffness and Adhesion in Spinal Cord Tumor Using Magnetic Resonance Elastography
Brief Title: MRE Evaluation for Spinal Cord Tumor Surgery: Stiffness and Adhesion Assessment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Yu Shi, Deputy director of department of radology, Shengjing Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ShengjingH_brain2023
Record Dates: First submitted 2023-07-15; First posted 2023-07-24 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Spinal Cord Tumors
Keywords: MRE; Slip Interface Imaging; Glioma; Magnetic Resonance Elastography; Spinal meningioma; Neurofibroma; Ependymoma; Astrocytoma; Glioblastoma; Spinal lipoma
MeSH Terms: conditions — Spinal Cord Neoplasms; Glioma; Meningioma; Neurofibroma; Ependymoma; Astrocytoma; Glioblastoma | interventions — Elasticity Imaging Techniques; Restraint, Physical

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic（MRE, tumor grading of stiffness and adhesion） (Experimental): Patients undergo a preoperative routine MRI scan and MRE the day before their scheduled surgery. During surgery, the tumor stiffness and adhesion are assessed and recorded by the surgeon according to established evaluation criteria. It is important to note that the surgeon does not have prior knowledge of the tumor's specific stiffness and adhesion before the surgery. This information is typically obtained through intraoperative assessment and observation.
  Interventions: Diagnostic Test: Magnetic Resonance Elastography; Procedure: Assessment and Recording

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Elastography — Undergo MRE and routine MRI
  Other Names: MRE
Procedure: Assessment and Recording — Undergo grading and recording of tumor stiffness and adhesion during surgery

SUMMARY:
In spinal cord tumors requiring surgical intervention, the resection difficulty is determined by two significant factors: tumor stiffness and adhesion to surrounding tissue.

The stiffness of the tumor dictates the complexity of removal, while strong adhesion presents additional challenges during the surgical procedure.

This clinical trial aims to assess the clinical utility of magnetic resonance elastography (MRE), in evaluating the stiffness and adhesion of spinal cord tumors and guiding surgical planning to selecting the most appropriate surgical approach for patients with spinal cord tumors.

DETAILED DESCRIPTION:
Spinal cord tumors are a common condition in neurosurgery, including neurofibroma, spinal meningioma, ependymoma, glioma, spinal lipoma, and so on.

Magnetic resonance imaging (MRI) plays a crucial role in the preoperative evaluation and planning of spinal cord tumor surgery. It provides detailed information about the tumor's location, size, and relationship to adjacent structures.

However, routine MRI may not always provide sufficient information about the tumor's stiffness or adhesion, which can impact surgical planning and postoperative outcomes. Magnetic resonance elastography and slip interface imaging can help measure the mechanical properties of tissues, including their stiffness or adhesion.

By combining the above methods, surgeons can identify areas of potential tumor adherence or invasion into surrounding structures, allowing for more precise surgical resection and minimizing the risk of damage to critical neural tissue.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing spinal cord tumor resection surgery are eligible for inclusion in the study cohort.

Exclusion Criteria:

* Patients with metallic implants or foreign bodies in their bodies (pacemakers, artificial metallic heart valves, metal joints, metal implants, and those who cannot remove dentures, insulin pumps, or contraceptive rings)
* Pregnant women in the first trimester (within three months)
* Patients with severe claustrophobia or anxiety
* Patients with severe fever
* Patients who can not tolerate MRE
* Patients with vascular malformations and aneurysms.
* Patients who do not sign an informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Surgical assessment of tumor stiffness | Baseline to 6 weeks
  The surgeon will score the tumor stiffness in seven aspects, ranging from 1 to 5 points: Tumor size; Shape of tumor; Tumor texture; Stiffness of the tumor's capsule; Stiffness of the tumor's central region; Primary methods of tumor removal; Features of tumor's capsule.
Surgical assessment of tumor adhesion | Baseline to 6 weeks
  The surgeon will score the tumor's adhesion based on seven aspects, ranging from 1 to 4 points: Stripping instruments; Frequency of use of sharp instruments; Adhesion range; Degree of tumor resection; Cranial nerve anatomy preservation; Brain tissue anatomy preservation; Neurological function (compared with preoperative).

CONTACTS AND LOCATIONS:
Overall Officials: Yu Shi, MD, Principal Investigator — Shengjing Hospital; Anhua Wu, MD, Principal Investigator — Shengjing Hospital; Wen Cheng, MD, Principal Investigator — Shengjing Hospital
Locations (1):
- Shengjing Hospital, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Murphy MC, Huston J 3rd, Glaser KJ, Manduca A, Meyer FB, Lanzino G, Morris JM, Felmlee JP, Ehman RL. Preoperative assessment of meningioma stiffness using magnetic resonance elastography. J Neurosurg. 2013 Mar;118(3):643-8. doi: 10.3171/2012.9.JNS12519. Epub 2012 Oct 19. PMID 23082888
- [Background] Hughes JD, Fattahi N, Van Gompel J, Arani A, Meyer F, Lanzino G, Link MJ, Ehman R, Huston J. Higher-Resolution Magnetic Resonance Elastography in Meningiomas to Determine Intratumoral Consistency. Neurosurgery. 2015 Oct;77(4):653-8; discussion 658-9. doi: 10.1227/NEU.0000000000000892. PMID 26197204
- [Background] Yin Z, Lu X, Cohen Cohen S, Sui Y, Manduca A, Van Gompel JJ, Ehman RL, Huston J 3rd. A new method for quantification and 3D visualization of brain tumor adhesion using slip interface imaging in patients with meningiomas. Eur Radiol. 2021 Aug;31(8):5554-5564. doi: 10.1007/s00330-021-07918-6. Epub 2021 Apr 14. PMID 33852045
- [Background] Yin Z, Hughes JD, Trzasko JD, Glaser KJ, Manduca A, Van Gompel J, Link MJ, Romano A, Ehman RL, Huston J 3rd. Slip interface imaging based on MR-elastography preoperatively predicts meningioma-brain adhesion. J Magn Reson Imaging. 2017 Oct;46(4):1007-1016. doi: 10.1002/jmri.25623. Epub 2017 Feb 14. PMID 28194925